CLINICAL TRIAL: NCT06583798
Title: Anatomical And Visual Outcomes of Retinal Re-surgeries in Silicone Oil Filled Eyes
Brief Title: Outcomes of Retinal Re-surgeries in Silicone Oil Filled Eyes
Acronym: ReSxinSO
Status: Completed | Type: Observational
Sponsor: Ahalia Foundation Eye Hospital (Other)
Responsible Party: Principal Investigator, Dr. Saurav Mahajan, Principal Investigator, Clinical Professor Adjunct, Ahalia Foundation Eye Hospital
Other Study IDs: 202201.; U1111-1312-4448 (Other: WHO UTN); TP232602676 (Other: NBEMS THESIS CONDUCT SECTION)
Record Dates: First submitted 2024-08-24; First posted 2024-09-04 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Retinal Detachment; Proliferative Vitreo-Retinopathy; Proliferative Diabetic Retinopathy
Keywords: Retinal Re-detachment; In silicone filled eyes; Under silicone oil; Proliferative Vitreoretinopathy
MeSH Terms: conditions — Retinal Detachment; Vitreoretinopathy, Proliferative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Resurgery In Silicone Oil Filled Eyes — * Alcon Luxor Biomicroscope with Non-contact BIOM (binocular indirect ophthalmomicroscope) viewing system was used.
  * 2 ports were made in Pars plana.
  * Top up of Silicone oil was done whenever needed.
  * Membrane peeling with relaxing retinectomy / drainage retinotomy, haemostasis and endolaser were done under Silicone oil as required.
  * After the re surgery, the patients were advised to maintain prone position.

SUMMARY:
Anatomical and Visual outcomes of retinal re-surgeries done in silicone oil filled eyes

DETAILED DESCRIPTION:
* Basic demographic profile including Name, Age, Gender, Place of Residence will be documented.
* structured questionnaire will be used to collect information regarding systemic diseases including Diabetes mellitus and its duration, Hypertension, Dyslipidemia , any cardiovascular diseases, any history of ocular trauma or any other ocular comorbidities.
* Details of the primary retinal surgery including indication, date of surgery, Name of the procedure will be noted
* Details of re surgery including indication (retinal pathology), timing of the re surgery from the primary surgery, preoperative Best Corrected Visual Acuity(BCVA) A using log MAR (Minimum Angle of resolution)) chart at 3 meters, intra ocular pressure using non contact Reichert 7 tonometry will be noted.
* Slit lamp bio-microscopy of the anterior segment using Topcon slit lamp biomicroscope,90 Diopter lens examination and indirect ophthalmoscopy with 20 Diopter lens of the fundus will be done.
* Spectral domain OCT(Optical coherence Tomography) with Zeiss Cirrus HD OCT (High Definition- Optical Coherence tomography) machine will be done for documentation of the status of macula in whichever cases possible.
* Re surgery will be done by a single Senior consultant in all the cases. Alcon Luxor Biomicroscope with Non contact BIOM (binocular indirect ophthalmomicroscope ) viewing system will be used. 2 ports will be made. Top up of Silicone oil will be done whenever needed. Membrane peeling with relaxing retinectomy / drainage retinotomy , haemostasis and endolaser will be done under Silicone oil as required. After the re surgery, the patient will be advised to maintain prone position.
* After the re surgery the BCVA(Best Corrected Visual Acuity), IOP (Intraocular pressure) will be noted on first visit at 15 days, 3rd month and 6th month follow up.
* Fundus examination will be done at all visits. Spectral Domain OCT(Optical coherence Tomography) will be done at all visits to see the status of macula.

STATISTICAL ANALYSIS

* Data entry will be done in Microsoft excel and analysed using the latest SPSS (Statistical Package for the Social Sciences) software.
* Wherever required, descriptive analysis will be done
* Chi square test will be used to find the statistical significance among the qualitative data, •two-tail t test will be used to find statistical significance among the quantitative data pre and post operatively.
* Other statistical tests will be used depending upon the need for post hoc analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had under gone the primary retina surgery at Ahalia Foundation Eye Hospital / elsewhere for retinal detachment secondary to various retinal pathologies and underwent re surgery during their follow up at Ahalia Foundation Eye Hospital during the study period.
* Patients whose proper follow up to 6 months after re surgery were maintained during the study period.
* No history of any additional eye disease other than h/o cataract surgery or primary RD repair.
* Patients who were willing to be a part of the study and willing to provide informed written consent.

Exclusion Criteria:

* Patients who did not come for any of the follow up included in the study.
* Patients who had history of ocular trauma after the primary surgery.
* Patients who have any other ocular comorbidities other than cataract.
* Patients who had undergone multiple previous re surgeries for retinal detachment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (South Indian Population) who attended retina Out patient department in Ahalia Foundation Eye Hospital, Palakkad and had to undergo Resurgery for Retinal Redetachment in various retinal pathologies
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Best Corrected Visual Acuity as assessed by LogMAR (Logarithm Minimum Angle of Resolution) chart | 6 months after Resurgery; 1 month post Silicone oil removal in eyes undergoing silicone oil removal
  * Change in mean Best Corrected Visual Acuity from Pre-operative time to 6 months post Re-surgery in silicone oil filled eyes
  * Change in mean Best Corrected Visual Acuity from Pre-operative time to 6 months post Re-surgery in silicone oil filled eyes with primary diagnosis of Diabetic Macular Tractional detachment
  * Change in mean Best Corrected Visual Acuity from Pre-operative time to 6 months post Re-surgery in silicone oil filled eyes with primary diagnosis of Rhegmatogenous retinal detachment
  * Change in mean Best Corrected Visual Acuity from Pre-operative time to 1month post Silicone oil Removal in eyes undergoing Silicone oil removal after Re-surgery in silicone oil filled eyes
Number and Percentage of eyes with Retina Reattched after resurgery in Silicone oil filled eyes | •6 months post resurgery; •3 months post silicone oil removal in Patients who underwent silicone oil removal
  * Total Number and Percentage of eyes with Retina Re-attached after re-surgery in Silicone oil filled eyes
  * Number and Percentage of eyes with Retina Re-attached after re-surgery in Silicone oil filled eyes having primary diagnosis of Diabetic Macular Tractional Detachment
  * Number and Percentage of eyes with Retina Re-attached after re-surgery in Silicone oil filled eyes having primary diagnosis of Rhegmatogenous retinal Detachment
  * Number and Percentage of eyes after re-surgery in Silicone oil filled eyes who underwent Silicone oil removal later
  * Number and Percentage of eyes who had retinal re-detachment after undergoing Silicone oil removal later

SECONDARY OUTCOMES:
number and percentage of patients having Best Corrected Visual Acuity of 1.6 Log Units | 6 months
  • number and percentage of patients having Best Corrected Visual Acuity of 1.6 Log Units or better pre-operatively and 6 months after re-surgery in silicone oil filled eyes
Number and percentage of eyes/patients having various risk factors for retinal detachment after primary surgery in silicone oil filled eyes | 6 months
  * Number and percentage of eyes having Proliferative Vitreoretinopathy under silicone oil
  * Number and percentage of eyes having retinal breaks under silicone oil
  * Number and percentage of patients having Epimacular membranes under silicone oil
  * Number and percentage of patients having associated systemic comorbities- diabetes, hypertension, cardiac issues, dyslipidemia, chronic kidney disease
Number and percentage of eyes/patients with adverse events intraoperative and post re-surgery in silicone oil filled eyes | 6 months post resurgery; 3 months post Silicone oil removal
  * Number and percentage of eyes with cataract progression post re-surgery in silicone oil filled eyes
  * Number and percentage of patients who underwent concurrent cataract surgery along with re-surgery in silicone oil filled eyes
  * Number and percentage of eyes with Epiretinal membrane post re-surgery in silicone oil filled eyes
  * Number and percentage of eyes with Silicone oil migration to Anterior chamber post re-surgery in silicone oil filled eyes
  * Number and percentage of patients with Corneal decompensation post re-surgery in silicone oil filled eyes
  * Number and percentage of patients with Retinal re-detachment post Silicone oil removal
  * Number and percentage of patients with Postoperative hypotony post Silicone oil removal
IOP change post Retinal Resurgery in silicone oil filled eyes | 6 months
  •Change in mean IOP before and after re-surgery in silicone oil filled eyes

CONTACTS AND LOCATIONS:
Overall Officials: Rajkumar Maheshwari, MS, Principal Investigator — Ahalia Foundation Eye Hospital; C R Asla Jahan, DNB, Principal Investigator — Ahalia Foundation Eye Hospital; Saurav Mahajan, MS, Principal Investigator — Ahalia Foundation Eye Hospital
Locations (1):
- Ahaliafoundation Eye Hospital, Palakkad, Kerala, India

IPD SHARING:
Plan to Share IPD: No